CLINICAL TRIAL: NCT00745719
Title: A Pilot Study to Evaluate the Efficacy of Total Parathyroidectomy in Retarding Cardiovascular Calcification in End-stage Renal Disease Patients
Brief Title: Parathyroidectomy in Endstage Renal Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Dr. Angela Yee-Moon Wang, Honorary Associate Professor, The University of Hong Kong
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: A111-102
Record Dates: First submitted 2008-09-01; First posted 2008-09-03 (Estimated); Last update posted 2020-08-05 (Actual); Status verified 2020-08

CONDITIONS: Endstage Renal Disease
Keywords: parathyroidectomy; cardiovascular; bone; endstage renal disease
MeSH Terms: interventions — Parathyroidectomy

STUDY DESIGN:
Intervention Model Description: Parathyroidectomy group versus natural disease control group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 1 (Experimental): surgical total parathyroidectomy with forearm autografting
  Interventions: Procedure: parathyroidectomy

INTERVENTIONS:
Procedure: parathyroidectomy — total parathyroidectomy with forearm autografting
  Other Names: total parathyroidectomy with forearm autografting

SUMMARY:
To test the hypothesis that total parathyroidectomy retards cardiovascular calcification, improves bone mineral density, reduces cardiac hypertrophy and arterial stiffening in end-stage renal disease patients on maintenance dialysis.

DETAILED DESCRIPTION:
Secondary hyperparathyroidism (SHPT) in patients with end-stage renal disease contributes to increased cardiovascular morbidity and mortality via different mechanisms. Uncontrolled hyperparathyroidism is associated with left ventricular hypertrophy and has been implicated in the development of cardiac interstitial fibrosis and diastolic dysfunction.

ELIGIBILITY:
Inclusion Criteria:

* Endstage renal disease patients receiving either long-term hemodialysis or peritoneal dialysis treatment, with elevated intact parathyroid hormone (iPTH) levels > 500pg/ml on two or more occasions.
* Patients with parathyroid nodular or diffuse hyperplasia identified by ultrasound imaging or radioisotope scan.
* Patients who provide informed consent for the study.

Exclusion Criteria:

* Patients with significant background valvular heart disease
* Patients who are unfit for general anaesthesia
* Patients with acute myocardial infarction within recent two months
* Patients with poor general condition
* Patients with plans for living related kidney transplant within 1 year
* Patients with previous history of parathyroidectomy
* Patients with calciphylaxis
* Patients with underlying active malignancy
* Patients with contraindication for MRI

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 122 (Actual)
Dates: Start 2007-03; Primary Completion 2011-09 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Change in vascular and valvular calcium scores | 12 months

SECONDARY OUTCOMES:
Change in bone mineral density | 12 months
change in aortic pulse wave velocity, | 12 months
change in left ventricular mass, volume and function | 12 months
changes in quality of life scores | 12 months
changes in iPTH | 6 and 12 months
changes in Serum calcium and phosphate | 6 and 12 months
changes in alkaline phosphatase | 6 and 12 months
changes in handgrip strength | 12 months
changes in subjective global assessment | 6 and 12 months
changes in serum albumin | 6 and 12 months
changes in inflammatory marker | 12 months
changes in HOMA index | 6 and 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Angela YM Wang, MD, PhD, Principal Investigator — Queen Mary Hospital, University of Hong Kong
Locations (1):
- Queen Mary Hospital, Tung Wah Hospital, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No